CLINICAL TRIAL: NCT06348914
Title: Knowledge of Vital Pulp Therapy in Permanent Teeth Among a Group of Dental Students in Egypt: A Cross-sectional Study.
Brief Title: Knowledge of Vital Pulp Therapy in Permanent Teeth Among a Group of Dental Students in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Maher Gindy, Resident in pediatric dentistry department at Misr International University, Cairo University
Other Study IDs: 6991
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Vital Pulp Therapy
Keywords: Vital Pulp Therapy; VPT; Permanent teeth; Dental Students; Egypt

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Knowledge assessment — survey on knowledge of a group of dental students regarding vital pulp therapy
Other: Educational Material — An awareness lecture on vital pulp therapy will be given to a group of the students right after they answer the questionnaire for the first time.

SUMMARY:
Conducting this questionnaire will help in collecting information about the extent of knowledge of vital pulp therapy in permanent teeth among dental students in Egypt. This will aid in identifying the knowledge gap, interest, and challenges regarding utilization of vital pulp therapy in permanent teeth.

ELIGIBILITY:
Inclusion Criteria:

* Dental students who live in Egypt.
* Dental students who are willing to participate
* Fifth-year students.

Exclusion Criteria:

-Responses with incomplete information

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A group of dental students in Egypt
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2024-11-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge of vital pulp therapy | from the 10th of September 2024 to the 10th of October 2024
  Measured by a questionnaire, and the measuring unit is multiple choice questions.

SECONDARY OUTCOMES:
Knowledge after awareness about vital pulp therapy | from the 10th of October 2024 to the 10th of November 2024
  Measured by a questionnaire, and the measuring unit is multiple choice questions.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] AAE Position Statement on Vital Pulp Therapy. J Endod. 2021 Sep;47(9):1340-1344. doi: 10.1016/j.joen.2021.07.015. Epub 2021 Aug 3. No abstract available. PMID 34352305
- [Background] American Academy of Pediatric Dentistry. Pulp therapy for primary and immature permanent teeth. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2022:415-23
- [Background] Bogen G, Dammaschke T, Chandler N. Vital pulp therapy. In: Berman L, Hargreaves KM, editors. Pathways of the Pulp. 12th ed. St. Louis, MO: Elsevier; 2021.
- [Background] Guan X, Zhou Y, Yang Q, Zhu T, Chen X, Deng S, Zhang D. Vital Pulp Therapy in Permanent Teeth with Irreversible Pulpitis Caused by Caries: A Prospective Cohort Study. J Pers Med. 2021 Nov 1;11(11):1125. doi: 10.3390/jpm11111125. PMID 34834477
- [Background] Parmar G, Singh S, Hegde JA, Kumar M, Kalyan S. Launching a new fellowship in microrestorative and endodontics for postgraduates in conservative dentistry and endodontics. J Conserv Dent. 2020 Jul-Aug;23(4):370-373. doi: 10.4103/JCD.JCD_328_20. Epub 2021 Jan 16. PMID 33623238
- [Background] Wisniewski JF, Norooz S, Callahan D, Mohajeri A. Survey of Vital Pulp Therapy Treatment in Permanent Dentition Being Taught at U.S. Dental Schools. J Endod. 2022 Sep;48(9):1107-1112. doi: 10.1016/j.joen.2022.06.009. Epub 2022 Jul 5. PMID 35798124
- [Background] Kakudate N, Yokoyama Y, Sumida F, Matsumoto Y, Gordan VV, Gilbert GH. Dentists' practice patterns of treatment for deep occlusal caries: Findings from a dental practice-based research network. J Dent. 2019 May;84:76-80. doi: 10.1016/j.jdent.2019.03.009. Epub 2019 Mar 29. PMID 30935965
- [Background] Doumani MD, Arnous WA, Alsafadi MF, Alnazer HA, Alanazi SM, Alotaibi KS, Al-Ammari AI. The Vital Pulp Therapy of Permanent Teeth: A Dental Practitioner's Perspective from Saudi Arabia. J Int Soc Prev Community Dent. 2020 Jun 15;10(3):300-308. doi: 10.4103/jispcd.JISPCD_69_19. eCollection 2020 May-Jun. PMID 32802776